CLINICAL TRIAL: NCT00275964
Title: Development of Active Safety Surveillance System for Traditional Chinese Medicine
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health (Ambiguous)
Other Study IDs: 920807
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2005-06

CONDITIONS: Climacteric Symptoms; Hot Flushes and/or Sweats

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: TMN-1

SUMMARY:
Context:Clinical trials demonstrating increased risk of cardiovascular disease and breast cancer among women randomized to hormone replacement therapy have attracted people's focus on the alternative therapy for menopausal symptoms. This study drug- a mixture of CHIA-WEI-HSIAO-YAO-SAN, CHIH-PO-TI-HUANG-WAN, HSIANG-SHA-LIU-CHUN-TZU-TANG (TMN1) is widely used as an alternative to hormonal therapies for hot flush in Taiwan. However, there is a paucity of data supporting their efficacy and safety.

Objective:To evaluate the safety and efficacy of TMN1 in the treatment of hot flush.

Design and Setting:A multi-center, prospective, observational follow-up study was conducted from July 2003 to December 2004 in 4 hospitals.

Participants:In total, 136 eligible subjects entered this study. They were required to take study drug 3 times a day for 12 weeks and make 9 visits at scheduled time for follow up efficacy and safety evaluations.

Main Outcome Measures:During the observation period, the investigators and study nurses actively enquired subjects if there was any adverse event (AEs) occurring to them by using Traditional Chinese medicine Adverse Events (TCM AE) questionnaire which includes 20 AEs proposed by experienced CM doctors as most commonly seen in the use of study drug. Every subject's complaint or abnormal laboratory value were carefully examined for possible causality and reviewed and decided by the research team. The primary outcome measure was the mean changes from baseline to week 12 in terms of frequency of hot flush and the severity of menopausal symptoms measured by the Kupperman Menopause Index. The secondary outcome measures included changes in quality of life measured by World Health Organization Quality of Life (WHOQOL) questionnaire, and adverse events monitored actively by a global assessment of tolerability. During the study period, every subject also received tests on routine hematology, biochemical function, and gynecologically relevant hormones at baseline visit, 4 weeks and 12 weeks after medication.

ELIGIBILITY:
Inclusion Criteria:

1. women between age of 45 and 55 and suffered from hot flushes and/or sweats
2. had not participated in any trial within the previous 3 months before beginning this study
3. were willing to participate in the trial and give written informed consent

Exclusion Criteria:

1. had received any form of hormonal therapy within 3 months prior to the study
2. had been diagnosed with any form of cancer and under treatment
3. were afflicted with abnormal uterine bleeding and unknown etiology
4. had hypertension or diabetes mellitus and were under treatment for these conditions
5. had any abnormal finding for kidney, liver, or thyroid functions
6. were currently taking antidepressants, alpha or beta-blocking agent, e.g., clomidine, ergot, ergot derivatives, or anti-estrogen medications such as tamoxifen and/or herbal hormones (isoflavon
7. were suffering from arrhythmia or any other form of heart disease.

Ages: 45 Years to 55 Years | Sex: Female
Age Groups: Adult
Dates: Start 2004-02; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Jung Der Wang, M.D., Sc.D.,, Study Director — Institute of Occupational Medicine and Industrial Hygiene, National Taiwan University College of Public Health